CLINICAL TRIAL: NCT06813560
Title: Parental Stress and Attachment in Premature Infants in Their First Months of Life in Early Months of Life in Child Development and Early Care Centres.
Brief Title: Parental Stress and Attachment in Preterm Infants
Status: Not yet recruiting | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: FUNDACIÓN SALUD INFANTIL (Unknown)
Responsible Party: Principal Investigator, Jose Miguel Soria Lopez, Clinical Professor, Cardenal Herrera University
Other Study IDs: CEEI24/544
Record Dates: First submitted 2024-12-20; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Premature Birth; Psychological Stress; Physiological Stress
MeSH Terms: conditions — Premature Birth; Stress, Psychological | interventions — Galvanic Skin Response; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature mothers: mothers who have given birth before 37 weeks' gestation
  Interventions: Diagnostic Test: hair cortisol; Diagnostic Test: salivary cortisol; Diagnostic Test: salivary Oxytocin; Diagnostic Test: Bayley-III Child Development Assessment Scales; Diagnostic Test: Strange Situation; Diagnostic Test: Parenting Stress Index (PSI); Diagnostic Test: Perinatal Risk Inventory; Diagnostic Test: Neonatal Behavioural Assessment (NBAS); Diagnostic Test: Galvanic Response; Diagnostic Test: electrocardiography (ECG); Diagnostic Test: Breathing respiratory rate
- mothers with full-term births (control group): mothers who have given birth after 37 weeks gestation
  Interventions: Diagnostic Test: hair cortisol; Diagnostic Test: salivary cortisol; Diagnostic Test: salivary Oxytocin; Diagnostic Test: Bayley-III Child Development Assessment Scales; Diagnostic Test: Strange Situation; Diagnostic Test: Parenting Stress Index (PSI); Diagnostic Test: Perinatal Risk Inventory; Diagnostic Test: Neonatal Behavioural Assessment (NBAS); Diagnostic Test: Galvanic Response; Diagnostic Test: electrocardiography (ECG); Diagnostic Test: Breathing respiratory rate

INTERVENTIONS:
Diagnostic Test: hair cortisol — To extract cortisol from the hair, the sample is carefully sectioned into segment lengths that will approximate the time period of interest (from the outermost part, if the hair is 3 cm long, the cortisol secreted proportionally by the individual in the last 3 months of life will be extracted). Then, an approximate average weight per sample of 150 mg will be selected. The samples will be individualised and placed in eppendorfs (one for each patient) and sprayed with scissors. After incubation in methanol for 36 hours, the supernatant portion is extracted, which already contains dissolved cortisol. This solution shall be evaporated to dryness, and then the pellet shall be reconstituted with phosphate (PBS). A commercial kit for the quantification of cortisol by immunoassay (ELISA Victor X5) shall be used. The ELISA kit for the detection of cortisol in saliva (ELISA Kits ' Cortisol ELISA Kits Human Cortisol Competitive ELISA Kit ,Invitrogen).
Diagnostic Test: salivary cortisol — Three saliva samples will be collected from each subject, at 8:00, 15:00 and 23:00 hours. Before collecting the saliva they will be instructed to rinse their mouth with cold water, without brushing their teeth. They should also not eat or drink in the hour before the sample is taken. Approximately 1 ml of saliva, collected by direct expectoration into an ependymal tube, shall be obtained and the samples shall be stored for 24 hours at 4°C . Subsequently, samples shall be centrifuged at 2 500 rpm/10 min and the supernatant shall be stored at -20 °C until processing by ELISA kit as per the above protocol.
Diagnostic Test: salivary Oxytocin — The treatment and collection of saliva as a biological sample shall be identical to the protocol described for the determination of cortisol. The determination of oxytocin shall be carried out by the use of ELISA kit for immunoassay (Oxytocin ELISA Kit (ab133050 ABCAM)
Diagnostic Test: Bayley-III Child Development Assessment Scales — They are a set of three standardised assessment scales, which assess the cognitive, motor and language development of children aged 1 and 42 months. For our study, we will use only the motor scale, which is composed of two subscales, the gross motor scale and the fine motor scale. This motor scale is composed of 138 items (the gross motor scale is composed of 72 items and the fine motor scale of 66 items) which assess the degree of control of the body, the coordination of large muscle masses and the manipulative ability of hands and fingers. The total administration time of the motor area for 12-month-old children, as in the case of the sample, is between 15 and 20 minutes.
Diagnostic Test: Strange Situation — The Strange Situation is a standardised observational procedure in which the child is exposed to two moments of separation from his/her attachment figure, two moments of reunion with the attachment figure and moments in which he/she interacts with an unknown person, specifically 8 episodes (lasting 3 minutes) in which the level of stress provoked in the child increases in intensity as the situation progresses. It is estimated to last around 20 minutes. It is assessed on a 7-point Likert-type scale, so that low scores indicate low frequency and intensity of the behaviour. These responses allow us to identify three types of attachment: secure attachment, insecure-avoidant attachment and insecure-ambivalent attachment. The strange situation only allows us to assess attachment in children between 1 and 2 years of age.
Diagnostic Test: Parenting Stress Index (PSI) — It assesses the stress experienced in parenting through several subscales such as parental distress, dysfunctional parent-child interaction and whether the child is a difficult child based on how parents perceive their children's behaviour.
Diagnostic Test: Perinatal Risk Inventory — - The Perinatal Risk Inventory is a measuring instrument that provides information on the neonatal situation prior to discharge and facilitates an estimate of the biological risk that the child may present from a very early age. The factors that are analysed in this inventory are evaluated with a score from 0 to 3 for each of the factors mentioned above, ranging from a minimum of 0 points to a maximum of 51. The levels of risk were determined as follows:
  1. Low Neonatal Risk: 0 to 6 points.
  2. Moderate Neonatal Risk: 7 to 9 points.
  3. High Neonatal Risk: 10 or more points.
Diagnostic Test: Neonatal Behavioural Assessment (NBAS) — is an assessment technique that provides a profile of scores that allows us to detect a possible alteration or pathology, but at the same time, within normal parameters, to detect both the potential or 'strong points' and the problems or 'weak points' of the newborn, as well as their peculiar ways of acting and reacting to environmental variables. Therefore, a profile of the child's behavioural characteristics is obtained, which can be considered as a first outline of the child's temperamental traits. It evaluates the behavioural repertoire of the newborn in 28 behavioural items that are assessed according to a 9-point scale. The scale also includes an assessment of neurological status in 18 reflex items, each with a 4-point rating. In the second edition of the NBAS a series of 7 supplementary items were added with the intention of better capturing the degree of fragility and the quality of behaviour of high-risk children.
Diagnostic Test: Galvanic Response — Galvanic Response: has the function of measuring the galvanic response of the skin, also known as electrodermal activity (EDA). It is used to record the electrical behaviour of the skin, which varies according to the activity of the sweat glands. This measurement of electrodermal activity is essential for studying the activity of the autonomic nervous system, which controls involuntary body functions such as sweating and heart rate. It will be measured with the BIOPAC MP36R device.
Diagnostic Test: electrocardiography (ECG) — ECG is used as a monitoring target for various cardiovascular conditions. It will be measured with the BIOPAC MP36R device.
  P, Q, R, S, T, U waves; QRS complex, PR interval and QT interval and PR segment and ST segment.
Diagnostic Test: Breathing respiratory rate — The transducer is attached to a strap that is placed around the subject's chest, allowing chest movements to be detected during breathing. The strap ensures a secure and comfortable fit for the subject during the measurement process. This transducer is used in conjunction with other BIOPAC components to assess physiological responses. The data obtained from the transducer provides information on respiratory patterns and their relationship to other physiological measures. It will be measured with the BIOPAC MP36R device.

SUMMARY:
Introduction: Advances in neonatology mean a significant reduction in mortality in premature infants as well as an increase in the risk of morbidity in the medium, short and long term. Furthermore, previous studies have linked prematurity, as an associated risk factor, with possible alterations in the bonding between the child and his or her mother in the first years of life. The possible impact that the stay in the neonatal unit may have on the mental health of the parents is noted. In fact, several studies have shown that the hospital environment of neonatal units may contribute to increased stress and anxiety in mothers. On the other hand, prematurity is one of the causes of referral to Child Development and Early Care Centres, to address their development in the first years of life, as well as for family support. One of the functions of early childhood professionals is to guarantee the development of a secure attachment between the child and his or her caregivers. Little is known about whether maternal stress levels can influence mother-child interactions and thus influence the attachment relationship in the early years of life.

Objective: to analyse the association between mothers' stress level due to preterm birth and attendance at a Child Development and Early Care Centre and child development and patterns of mother-child interactions.

ELIGIBILITY:
Inclusion Criteria:

* Children born under 37 weeks of gestation,
* Parents of legal age and who have sufficient cognitive capacity to understand the informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Children admitted to the Neonatal Unit and who start treatment at the Child Development and Early Care Centre of the Fundación Salud Infantil de Elche (Alicante, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
salivary cortisol (nmol/L) | Pre-intervention / a year post-intervention
  ELISA Kits ' Cortisol ELISA Kits Human Cortisol Competitive ELISA Kit ,Invitrogen. Quantification of cortisol and oxytocin: RT-2100C microplate reader, which is a general-purpose microprocessor-controlled photometric system designed to read and calculate biomarker assay results (optic ivymen system)
hair cortisol (nmol/L) | Pre-intervention / a year post-intervention
  ELISA Kits ' Cortisol ELISA Kits Human Cortisol Competitive ELISA Kit ,Invitrogen. Quantification of cortisol and oxytocin: RT-2100C microplate reader, which is a general-purpose microprocessor-controlled photometric system designed to read and calculate biomarker assay results (optic ivymen system)
salivary oxytocin (units/ml) | Pre-intervention / a year post-intervention
  ELISA Kits ' Cortisol ELISA Kits Human Cortisol Competitive ELISA Kit ,Invitrogen. Quantification of cortisol and oxytocin: RT-2100C microplate reader, which is a general-purpose microprocessor-controlled photometric system designed to read and calculate biomarker assay results (optic ivymen system)
electrocardiography (mV) | Pre-intervention / a year post-intervention
  BIOPAC MP36R device: ECG: P, Q, R, S, T, U waves; QRS complex, PR interval and QT interval and PR segment and ST segment
galvanic response by means of Skin conductance (SC) micro-siemens or micro-omhios | Pre-intervention / a year post-intervention
  BIOPAC MP36R device
breathing rate (breaths per minute) | Pre-intervention / a year post-intervention
  BIOPAC MP36R device
Parenting Stres Index (PSI) | Pre-intervention / a year post-intervention
  PSI-SF is a 36-item, self-report measure of parenting stress. It includes three subscales: Parental Distress (PD; e.g, "I feel trapped by my responsibilities as a parent", "I feel lonely and without friends"), Parent-Child Dysfunctional Interaction (PCDI; e.g, "Sometimes I feel my child doesn't like me and doesn't want to be close to me", "When I do things for my child I get the feeling that my efforts are not appreciated" ), and Difficult Child (DC; e.g, "My child makes more demands on me than most children", "My child gets upset easily over the smallest thing"). Each subscale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree), with subscales scores ranging from 12 to 60. A Total score is calculated by summing the three subscales scores, ranging from 36 to 180. Scores of 90 or above may indicate a clinical level of stress. Cronbach's alpha coefficients of .91 for PSI-SF total score, and .87, .80, and .85 for PD, PCDI, and DC subscales.
Perinatal Risk Inventory | Pre-intervention / a year post-intervention
  It consists of a total of 18 risk factors such as 1) Apgar score; 2) electro-encephalogram; 3) non-metabolic seizures; 4) intraventricular haemorrhage; 5) hydrocephalus; 6) neurological findings (not for hydrocephalus or HIV); 7) gestational age at birth; 8) weight for gestational age; 9) dysmorphias; 10) assisted ventilation; 11) cranial growth (children hospitalised 6 or more weeks); 12) cranial growth (children hospitalised less than 3 weeks); 13) polycythaemia; 14) meningitis; 15) hypoglycaemia; 16) congenital infections; 17) hyperbilirubinaemia; and 18) associated medical problems (not central nervous system). These factors are assessed with a score from 0 to 3 for each of the above factors, ranging from a minimum of 0 points to a maximum of 51 points. Risk levels:
  1. Low Neonatal Risk: 0 to 6 points.
  2. Moderate Neonatal Risk: 7 to 9 points.
  3. High Neonatal Risk: 10 or more points.
Neonatal Behavioural Assessment (NBAS) | Pre-intervention / a year post-intervention
  It evaluates the behavioural repertoire of the newborn in 28 behavioural items that are assessed according to a 9-point scale. The scale also includes an assessment of neurological status in 18 reflex items, each with a 4-point rating. The NBAS can be used without any adaptations for full-term children and can be used until the end of the second month of life. With the addition of supplementary items it can also be used with apparently healthy preterm infants (less than 37 weeks gestation) and for them, depending on the degree of immaturity, application is possible up to 48 weeks post-conceptional age. <7 points: low, suggests newborn distress requiring intervention.
  7-9 points: normal. child in good health.
Bayley-III Child Development Assessment Scales | Pre-intervention / a year post-intervention
  They are a set of three standardised assessment scales, which evaluate the cognitive, motor and language development of children aged 1 and 42 months. We will use only the motor scale, which is composed of two subscales, the gross motor scale and the fine motor scale. This motor scale is composed of 138 items (the gross motor scale is composed of 72 items and the fine motor scale of 66 items) which assess the degree of control of the body, the coordination of large muscle masses and the manipulative ability of hands and fingers. The total administration time of the motor area for 12-month-old children, as in the case of the sample, is between 15 and 20 minutes. average motor score: 100; <85=mild impairment; <70=moderate-severe impairment
Ainsworth's test (Strange Situation) | Pre-intervention / a year post-intervention
  The Strange Situation is a standardised observational procedure in which the child is exposed to two moments of separation from his/her attachment figure, two moments of reunion with the attachment figure and moments in which he/she interacts with an unknown person, specifically 8 episodes (lasting 3 minutes) in which the level of stress provoked in the child increases in intensity as the situation progresses. It is estimated to last around 20 minutes. It is assessed on a 7-point Likert-type scale, so that low scores indicate low frequency and intensity of the behaviour. These responses allow us to identify three types of attachment: secure attachment, insecure-avoidant attachment and insecure-ambivalent attachment. The strange situation only allows us to assess attachment in children between 1 and 2 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU Cardenal Herrera, plaza Reyes Catolico 19, 03204 Elche (alicante ), Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT06813560/Prot_SAP_ICF_000.pdf